CLINICAL TRIAL: NCT03969030
Title: Peer-Educator-coordinated vs Nurse-coordinated ART Refill for Adolescents and Young Adults Living With HIV in Lesotho - a Cluster Randomized Clinical Trial (PEBRA Trial)
Brief Title: Peer-Educator-coordinated vs Nurse-coordinated ART Refill for Adolescents and Young Adults Living With HIV in Lesotho
Acronym: PEBRA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Amstutz Alain (Other)
Collaborators: International AIDS Society (CIPHER grant) (Unknown); Swiss Tropical & Public Health Institute (Other); SolidarMed (Other); Sentebale (Other); University of Basel (Other); University Hospital, Basel, Switzerland (Other); Swiss National Science Foundation (Other)
Responsible Party: Sponsor-Investigator, Amstutz Alain, MD, Swiss Tropical & Public Health Institute
Organization: Swiss Tropical & Public Health Institute (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 2019-10
Record Dates: First submitted 2019-05-09; First posted 2019-05-31 (Actual); Last update posted 2021-06-02 (Actual); Status verified 2021-05

CONDITIONS: HIV/AIDS
Keywords: HIV; Sub-Sahara Africa; Lesotho; Differentiated Service Delivery; Adolescents and young adults living with HIV; ART service; Preference-based
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Intervention Model Description: PEBRA study is a cluster randomized, open-label, superiority trial in a resource-limited setting
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Participants in the intervention clusters are offered the PEBRA model. In the PEBRA model the ART visit/refill is coordinated by the Peer-Educator (PE) according to the participants' preferences, using a tablet-based application, called PEBRApp. The preference assessment entails the following three domains of DSD:
  1. ART Refill
  2. SMS notifications
  3. Support In each of the domains, the participants' preferences will be assessed and the most feasible option will be selected. The PEBRApp not only helps the PE to assess each participants' preference, but also to keep track of the ART refill, and to ensure regular contact between the PE and the participant. The model includes key innovative options such as individualized automatic SMS notifications and decentralized ART delivery.
  Interventions: Other: PEBRA model
- Control (No Intervention): Participants in the control clusters are offered standard of care: ART visit/refill is coordinated by the nurse, is mostly clinic-based, not adapted to youth, and differentiated according to clinical values (i.e. if VL suppressed then option of ART Refill in a Community Adherence Club).

INTERVENTIONS:
Other: PEBRA model — The participants in the intervention clusters are offered the PEBRA model. In the PEBRA model the ART visit/refill is coordinated by the PE, as much as feasible according to the participants' preferences. Thus, the preferences of each participant are captured at enrolment and after a strict schedule thereafter. The PE conducts the preference assessment using a tablet-based application, called PEBRApp, accoring to a specific schedule. First, the participant will be asked his/her preference regarding different domains of DSD (see below) and this will be entered into the PEBRApp. Secondly, the chosen preferences are assessed regarding feasibility with specific questions, as not all preference options are available to everyone all the time. The preference assessment entails the following three domains of DSD:
  1. ART Refill
  2. SMS notifications
  3. Support
  Arms: Intervention

SUMMARY:
Sub-Saharan Africa (SSA) is home to 85% of the adolescents and young people living with HIV (AYPLHIV) globally and they are heavily affected by the HIV/AIDS epidemic: AYPLHIV in SSA are the only population group for whom HIV-related mortality continues to increase, and they have overall poorer outcomes than all other age groups. Lesotho with worldwide the second-highest HIV prevalence shows a viral suppression rate among AYPLHIV of only 49%.

In order to address the multiple barriers in the adolescent HIV care cascade and their unique needs, multicomponent packages of differentiated service delivery (DSD) are a promising approach.

In close collaboration with different local stakeholders, the researchers designed a DSD model specifically for AYPLHIV, called the PEBRA model. In the PEBRA model the peer-educator (PE) plays a pivotal role, by coordinating the ART refill/care according to the patient's preferences using a tablet-based application, called PEBRApp (https://github.com/chrisly-bear/PEBRApp). The PEBRApp helps the PE to assess each participant's preference, to adapt the ART refill according to these preferences in a feasible manner, to keep track of the ART refill, and to ensure regular contact between the PE and the participant. The model includes key innovative options such as individualized automatic SMS notifications and decentralized ART delivery.

The PEBRApp was developed with ❤️ by Technify Maseru, Lesotho (www.technifyls.com) & Christoph Schwizer Zurich, Switzerland (www.christophschwizer.ch).

DETAILED DESCRIPTION:
STUDY DESIGN

PEBRA study is a cluster randomized, open-label, superiority trial in a resource-limited setting. The rational for a cluster randomized design with health facilities as clusters, is the high risk of cross-contamination between the study arms if randomization would be done at individual level. The clusters (health facilities) will be randomized (randomly-varying block sizes, 1:1 allocation) into the 2 groups using a computer-generated randomization list, stratified by district and size of the AYPLHIV cohort of each facility (<15 vs ≥15). The study will be conducted at 20 health facilities in three districts of Lesotho (Leribe, Butha-Buthe, Mokhotlong).

OBJECTIVES

The overall objective of this study is to evaluate the feasibility and effectiveness of a DSD model ("PEBRA model") among AYPLHIV.

As primary objective this study seeks to assess the rate of viral suppression among AYPLHIV 12 months after enrolment between the intervention clusters, where AYPLHIV were offered the PEBRA model, and the control clusters, where AYPLHIV were offered standard of care.

Secondary objectives include a comparison of adherence to ART, the level of perceived quality of ART care and patient service satisfaction, engagement in care, viral suppression, lost-to-follow-up (LTFU), mortality, and transfer out between the intervention and control clusters. Further objectives include a cost-effectiveness evaluation and qualitative research regarding acceptance, scalability and feasibility of the DSD model.

QUALITATIVE RESEARCH

Besides above outlined qualitative research (QoL, QoC, longitudinal description of participants' preference assessments) the researchers will explore the acceptability of the PEBRA model in a) Focus Group Dis-cussions (FGD) with study participants from the intervention clusters, and b) key informant interviews (KII) with the main stakeholders (District Health Management Team and different health center staff). We plan to conduct at least 2 FGD (with about 5 study participants) per district and 3 KII per district, ac-cording to the concept of saturation. Data will be collected by trained facilitators using piloted interview questionnaires and discussion guides, in the local language (Sesotho). Qualitative data will be record-ed, transcribed, translated into English and coded and analyzed using the Framework Method. All participants in this qualitative research will be required to sign a separate consent form to participate and to be recorded. These consent forms and interview questionnaires will be submitted as an amendment to the ethics committee in Lesotho at a later stage.

COST-EFFECTIVENESS ANALYSIS AND SYSTEM IMPACT EVALUATION

The researchers will perform a system impact evaluation and cost-effectiveness analysis, in order to estimate the im-pact of the PEBRA model on health benefits and costs. First, we will assess the direct costs of the PEBRA model. Secondly, we will assess the cost-effectiveness of the PEBRA model. Thirdly, we will as-sess the economic burden of the PEBRA model to the study participants, i.e. including both direct costs and the opportunity costs of their time. The assessment of direct costs includes staff costs (PEs, clinic staff, VHWs), personnel training costs (especially for the PEs), the cost of equipment needed (PEBRApp, logistics), medical costs to the participant (medication, laboratory tests, consumables, etc.), and non-medical costs to the participant (i.e. cost of transportation to ART service). Data to assess pa-tient level costs will be collected from a randomly selected sub-sample of study participants from each cluster arm, using medical expenditure records and interviews. Cost outcomes will include:

i) The average cost to the service provider per patient achieving the primary endpoint at 12 months in each cluster arm ('per patient suppressed provider cost') ii) The average cost to the patient per patient achieving the primary endpoint at 12 months in each cluster arm ('per patient suppressed patient cost') iii) The annual cost per patient in each cluster arm ('per patient year cost') iv) The cost-effectiveness of the PEBRA model with respect to viral suppression and engage-ment in care Costs will be reported as means (incl. standard deviations) and medians (incl. interquartile range) in local currency and US dollar and International Dollar.

PREFERENCE AND FEASIBILITY ASSESSMENT

The researchers will systematically assess the following exploratory analyses regarding feasibility and youth ART service preference:

1. Youth ART service preferences: Longitudinal description of participants' preference assessments
2. Feasibility of youth ART service according to preferences: Percentage of ART service delivered according to participants' preferences
3. Differentiated Impact of the different support options on key study outcomes

PILOT TRIAL

PEBRA model will be piloted at one representative health facility in Butha-Buthe district, that will be pragmatically chosen in collaboration with the District Health Management Team. The pilot trial will be crucial to assess feasibility of the PEBRA model and the study procedures. The same procedures apply in the pilot trial as in the main trial, using the same consent process and baseline data collection. One PE will be specifically trained for the pilot. Recruitment for the pilot will be closed once 3-5 study participants are enrolled and follow-up will last for 2.5 months after having enrolled the last participant. All endpoints that are evaluable "at 3 months (range 2.5 - 3.5)" will be assessed and analyzed. The aim of the pilot trial is to give a first insight into PEBRA model and provide detailed information for the main trial.

ELIGIBILITY:
Eligibility - clusters

Inclusion criteria:

1. the cluster is a public or missionary health center from the study districts, that offers ART services
2. the cluster has at least one PE who is willing to participate and fulfills the following criteria:

   1. underwent the Sentebale Peer-Educator two-weeks training
   2. attended and successfully passed the study training assessment

Exclusion criteria:

1. health facility authority opposed to trial participation (verbal assent)
2. the health facility is a hospital
3. the health facility is situated in an area without cellphone signal

Eligibility - individuals

1. Individual is living with HIV and in care in a participating cluster
2. Individual is 15-24 years old (AYPLHIV)
3. Informed consent given
4. Declares to seek the next follow-up visit at the same health facility

Ages: 15 Years to 24 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 307 (Actual)
Dates: Start 2019-11-01 (Actual); Primary Completion 2021-04-30 (Actual); Study Completion 2021-04-30 (Actual)

PRIMARY OUTCOMES:
In care with documented viral suppression | 12 months (range: 9 - 15 months) after enrolment
  In care with documented viral suppression at 12 months, defined as the proportion of participants in care with a documented VL <20 copies/mL 12 months (range: 9 - 15 months) after enrolment out of all participants enrolled

SECONDARY OUTCOMES:
Adherence to ART at 3 months (range 2.5 - 3.5), 6 months (range 5 - 8) and 12 months (range 9 - 15) after enrolment | 3 months (range 2.5 - 3.5), 6 months (range 5 - 8) and 12 months (range 9 - 15) after enrolment
  Assessed by 4 different setting- and age-validated ART adherence questions:
  1. pill count: change in percentage
  2. "When was the last time you missed any medications?" (i) past week, ii) 1-2 weeks ago, iii) 3-4 weeks ago, iv) never): Dichotomous outcome missed doses vs. no missed doses in the past month
  3. "ART missed at two or more consecutive days within last month?" ("drug holiday" question)
  4. "How would you rate your adherence over the last month" (i) very poor, ii) poor, iii) fair, iv) good, v) very good, vi) excellent): Dichotomous outcome adherent vs non-adherent (anything less than 'excellent')
Quality of Life (QoL) at 6 months (range 5 - 8) and 12 months (range 9 - 15) after enrolment | 6 months (range 5 - 8) and 12 months (range 9 - 15) after enrolment
  Assessed by WHO QoL in PLHIV: WHO HIV QoL questionnaire (whoqol_hiv_bref questionnaire with 31 five-point Likert Scale items with categorical outcomes
Perceived quality of ART Care / patient service satisfaction at 6 months (range 5 - 8) and 12 months (range 9 - 15) after enrolment | 6 months (range 5 - 8) and 12 months (range 9 - 15) after enrolment
  Assessed by a setting-validated QoC and patient service satisfaction questionnaire (12 five-point Likert Scale items with categorical outcome) by an external data collector, not the peer-educator
Engagement in care at 6 months | 6 months (range 5 - 8) after enrolment
  Engagement in care at 6 months, defined as the proportion of participants engaged in care 6 months (range 5 - 8) after enrolment out of all participants enrolled
Alternative viral suppression at 12 months | 12 months (range 9 - 15) after enrolment
  Alternative viral suppression at 12 months, defined as the proportion of participants with a documented VL <1000 copies/mL 12 months (range 9 - 15) after enrolment out of all participants enrolled
Engagement in care at 12 months | 12 months (range 9 - 15) after enrolment
  Engagement in care at 12 months, defined as the proportion of participants engaged in care 12 months (range 9 - 15) after enrolment out of all participants enrolled
All-cause mortality | 6 months (range 5 - 8) and 12 months (range 9 - 15) after enrolment
  All-cause mortality at 6 and 12 months, defined as the proportion of participants dead 6 months (range 5 - 8) and 12 months (range 9 - 15) after enrolment, respectively, out of all participants enrolled
LTFU at 6 and 12 months | 6 months (range 5 - 8) and 12 months (range 9 - 15) after enrolment
  LTFU at 6 and 12 months, defined as the proportion of participants LTFU 6 months (range 5 - 8) and 12 months (range 9 - 15) after enrolment, respectively, out of all participants enrolled
Transfer out at 6 and 12 months | 6 months (range 5 - 8) and 12 months (range 9 - 15) after enrolment
  Transfer out at 6 and 12 months, defined as the proportion of participants who transferred out to any other health facility (than the initially attached one) with known outcome (documented proof of follow-up visit or laboratory test) 6 months (range 5 - 8) and 12 months (range 9 - 15) after enrolment, respectively, out of all participants enrolled

OTHER OUTCOMES:
Serious Adverse Events (SAE) | within 12 months after enrolment
  The proportion out of all participants experiencing a Serious Adverse Events (SAE) within 12 months after enrolment

CONTACTS AND LOCATIONS:
Overall Officials: Niklaus Labhardt, MD MIH, Study Chair — Swiss TPH & University Hospital Basel & University of Basel; Alain Amstutz, MD, Principal Investigator — Swiss TPH & University Hospital Basel & University of Basel; Mathebe Kopo, Study Director — SolidarMed; Jennifer Brown, MSc, Study Director — Swiss TPH & University of Basel; Nadine Bachmann, MSc, Study Director — Swiss TPH & University of Basel; Thabo Lejone, MIH, Study Director — SolidarMed; Lebohang Sao, MD, Study Director — DHMT BB; Tracy Glass, PhD, Study Director — Swiss TPH & University of Basel
Locations (20):
- Lesotho (20):
  - Boiketsiso HC, Butha-Buthe
  - Linakeng HC, Butha-Buthe
  - Makhunoane HC, Butha-Buthe
  - Motete HC, Butha-Buthe
  - Muela HC, Butha-Buthe
  - Ngoajane HC, Butha-Buthe
  - Rampai HC, Butha-Buthe
  - St. Paul HC, Butha-Buthe
  - St. Peters HC, Butha-Buthe
  - Tsime HC, Butha-Buthe
  - Ha Lejone HC, Hlotse
  - Pontmain, Hlotse
  - Libibing HC, Mokhotlong
  - Linakaneng HC, Mokhotlong
  - Malefiloane HC, Mokhotlong
  - Mapholaneng HC, Mokhotlong
  - Moeketsane HC, Mokhotlong
  - Molikaliko HC, Mokhotlong
  - St. James HC, Mokhotlong
  - St. Martins HC, Mokhotlong

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, ICF
Time Frame: Any time.
Access Criteria: Data from this study, including deidentified participant data, study protocol, and informed consent documents will be made available to researchers. To access data, researchers should contact the corresponding author. Researchers will need to present a concept sheet for their proposed analysis. This will have to be reviewed and approved by all co-authors. The co-authors will consider overlap of the proposed project with active or planned analyses and the appropriateness of study data for the proposed analysis.

REFERENCES:
- [Derived] Seiler O, Kopo M, Kao M, Lejone TI, Tschumi N, Glass TR, Brown JA, Labhardt ND, Amstutz A. HIV Care Preferences among Young People Living with HIV in Lesotho: A Secondary Data Analysis of the PEBRA Cluster Randomized Trial. AIDS Res Treat. 2023 Apr 14;2023:8124192. doi: 10.1155/2023/8124192. eCollection 2023. PMID 39691584
- [Derived] Kopo M, Lejone TI, Tschumi N, Glass TR, Kao M, Brown JA, Seiler O, Muhairwe J, Moletsane N, Labhardt ND, Amstutz A. Effectiveness of a peer educator-coordinated preference-based differentiated service delivery model on viral suppression among young people living with HIV in Lesotho: The PEBRA cluster-randomized trial. PLoS Med. 2023 Jan 3;20(1):e1004150. doi: 10.1371/journal.pmed.1004150. eCollection 2023 Jan. PMID 36595523
- [Derived] Lejone TI, Kopo M, Bachmann N, Brown JA, Glass TR, Muhairwe J, Matsela T, Scherrer R, Chere L, Namane T, Labhardt ND, Amstutz A. PEBRA trial - effect of a peer-educator coordinated preference-based ART service delivery model on viral suppression among adolescents and young adults living with HIV: protocol of a cluster-randomized clinical trial in rural Lesotho. BMC Public Health. 2020 Mar 30;20(1):425. doi: 10.1186/s12889-020-08535-6. PMID 32228531
- See also: PEBRApp — https://github.com/chrisly-bear/PEBRApp

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-05-24): https://cdn.clinicaltrials.gov/large-docs/30/NCT03969030/Prot_SAP_000.pdf